CLINICAL TRIAL: NCT00001967
Title: Immunologic and Virologic Studies of Intermittent Versus Continuous HAART in the Treatment of HIV Disease
Brief Title: Intermittent Versus Continuous Medication in the Treatment of HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000020; 00-I-0020; NCT00001134 (obsolete NCT alias)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-11

CONDITIONS: HIV Infection
Keywords: HIV; HAART; Immunity; Toxicity; Resistance; Treatment Interruption
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

INTERVENTIONS:
Drug: HAART

SUMMARY:
Although highly active antiretroviral therapy (HAART) has been successful in suppressing plasma HIV RNA levels in infected patients, it has not resulted in eradication of virus. It is now clear that virus replication persists despite undetectable plasma viremia in individuals receiving HAART. In this regard, withdrawing HAART, even after prolonged periods of virus suppression, leads to an almost universal rapid rebound of plasma viremia. It is also now clear that prolonged, continuous HAART carries a risk of significant toxicity and side effects. These recent observations may argue for a different approach to HAART with the goals of: 1) durable suppression of virus replication, without an attempt at eradication, and 2) minimization of toxicity and side effects and improvement in patient life-style. Therefore, we propose to study the virologic and immunologic effects of intermittent versus continuous HAART in HIV-infected individuals as a possible means to achieve these goals. The primary protocol, Cohort 1, will be a randomized controlled study of 35 individuals receiving continuous HAART and 35 individuals receiving intermittent HAART with intervals of one month off therapy followed by two months on therapy. A second cohort of 10 individuals will serve as a pilot of 2 arms of 5 patients each to evaluate the potential of shorter on-off cycles to maintain suppression of plasma virus and boost HIV-specific immune responses. An extension of Cohort 2 will add 5 patients to the 7 days on/7 days off HAART arm with modified exclusion criteria and procedure schedule. We will analyze CD4+ T-cell counts, viral load, incidence of toxicity and side effects, HIV-specific immune responses and viral resistance to therapy and characterize the virus during rebound plasma viremia.

DETAILED DESCRIPTION:
Although highly active antiretroviral therapy (HAART) has been successful in suppressing plasma HIV RNA levels in infected patients, it has not resulted in eradication of virus. It is now clear that virus replication persists despite undetectable plasma viremia in individuals receiving HAART. In this regard, withdrawing HAART, even after prolonged periods of virus suppression, leads to an almost universal rapid rebound of plasma viremia. It is also now clear that prolonged, continuous HAART carries a risk of significant toxicity and side effects. These recent observations may argue for a different approach to HAART with the goals of: 1) durable suppression of virus replication, without an attempt at eradication, and; 2) minimization of toxicity and side effects and improvement in patient life-style. Therefore, we propose to study the virologic and immunologic effects of intermittent versus continuous HAART in HIV-infected individuals as a possible means to achieve these goals. The primary protocol, Cohort 1, will be a randomized controlled study of 45 individuals receiving continuous HAART and 45 individuals receiving intermittent HAART with intervals of one month off therapy followed by two months on therapy. A second cohort of 10 individuals will serve as a pilot study of 2 arms of 5 patients each to evaluate the potential of shorter on-off cycles to maintain suppression of plasma virus and boost HIV-specific immune responses. An extension of Cohort 2 will add 5 patients to the 7 days on/ 7 days off HAART arm with modified exclusion criteria and procedure schedule. Cohort 3 will be a pilot study of 5 individuals who will received 4 days off HAART followed by 3 days on HAART. Cohort 4 will be a pilot study of 8 individuals who will receive a once-daily HAART regimen administered as short cycle intermittent therapy of 7 days off drugs followed by 7 days on drugs. Cohort 5 will be a pilot study of 5 individuals who will receive 3 days off HAART followed by 4 days on HAART. We will analyze CD4+ T-cell counts, viral load, incidence of toxicity and side effects, HIV-specific immune responses and viral resistance to therapy and characterize the virus during rebound plasma viremia.

ELIGIBILITY:
INCLUSION CRITERIA:

Documentation of HIV-1 infection by licensed ELISA test kit and confirmed by a second method (e.g. Western Blot).

Absolute CD4+ T-cell count of greater than or equal to 300/mm(3) within 30 days before randomization (For patients who are status post-splenectomy, also CD4+ T-cell greater than 20%). For patients in cohort 2, the lowest documented CD4+ T-cell count must be greater than or equal to 200 cells/mm(3).

Receiving HAART (at least 2 NRTIs and an NNRTI or a PI) with at least 1 viral load test below the limit of detection (at least less than 500 copies/ml) greater than or equal to 3 months for cohort 1 and 4 and greater than or equal to 6 months for cohorts 2, 3 and 5 before screening.

A confirmatory viral load of less than 50 copies/ml prior to enrollment.

Age at least 18 years.

For women of childbearing potential, a negative pregnancy test (serum or urine) is required within 14 days prior to randomization.

Laboratory values (within 30 days prior to randomization):

AST no more than 5 times the upper limit of normal (ULN);

Total or direct bilirubin no more than 2 times the ULN unless there is a pattern consistent with Gilbert's syndrome or the patient is receiving indinavir;

Creatinine no more than 2.0 mg/dL;

Platelet count at least 50,000 microliters.

Willingness to provide blood samples for storage that may be used in future studies of HIV infection and/or immunopathogenesis.

EXCLUSION CRITERIA:

Concurrent malignancy, or any other disease state, requiring cytotoxic chemotherapy .

Symptomatic for significant HIV-related illnesses, such as opportunistic infections and malignancies other than mucocutaneous Kaposi's sarcoma .

Use of experimental antiretrovirals less than or equal to 6 months prior to enrollment. An exception may be made for hydroxyurea according to the judgment of the Principal Investigator.

For cohort 1 and the extension of cohort 2, current use of IL-2 or history of use of IL-2 . Cohorts 2, 3, 4 and 5, patients must not be currently receiving cycles of IL-2.

For the extension of cohort 2, participation in previous STI studies or off HAART for greater than 2 weeks consecutively in the last year.

Pregnancy or breastfeeding during the study period.

Significant cardiac, pulmonary, kidney, rheumatologic, gastrointestinal, or CNS disease as detectable on routine history, physical examination, or screening laboratory studies are excluded. If an abnormality is a contraindication to a specific drug, an alternative drug within the same class may be used.

Psychiatric illness that, in the opinion of the PI, might interfere with study compliance.

Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise patient safety.

Refusal to practice safe sex or use precautions against pregnancy (effective birth control or abstinence).

Known history or laboratory evidence of chronic hepatitis B infection including surface antigen positivity .

Patients not receiving salvage HAART, i.e. no evidence of clinical resistance to licensed antiretrovirals.

Patients in cohort 1 cannot be receiving nevirapine at the time of enrollment.

Patients receiving nevirapine or abacavir at time of enrollment.

Expanded access medications are not allowed at time of enrollment nor while on study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123
Dates: Start 1999-11; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Neumann AU, Tubiana R, Calvez V, Robert C, Li TS, Agut H, Autran B, Katlama C. HIV-1 rebound during interruption of highly active antiretroviral therapy has no deleterious effect on reinitiated treatment. Comet Study Group. AIDS. 1999 Apr 16;13(6):677-83. doi: 10.1097/00002030-199904160-00008. PMID 10397562
- [Background] Furtado MR, Callaway DS, Phair JP, Kunstman KJ, Stanton JL, Macken CA, Perelson AS, Wolinsky SM. Persistence of HIV-1 transcription in peripheral-blood mononuclear cells in patients receiving potent antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1614-22. doi: 10.1056/NEJM199905273402102. PMID 10341273
- [Background] Zhang L, Ramratnam B, Tenner-Racz K, He Y, Vesanen M, Lewin S, Talal A, Racz P, Perelson AS, Korber BT, Markowitz M, Ho DD. Quantifying residual HIV-1 replication in patients receiving combination antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1605-13. doi: 10.1056/NEJM199905273402101. PMID 10341272